CLINICAL TRIAL: NCT02306720
Title: An Observational, Longitudinal, Prospective, Long-Term Registry Of Patients With Hypophosphatasia (HPP)
Brief Title: Registry of Patients With Hypophosphatasia
Status: Enrolling by invitation | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-HPP-501
Record Dates: First submitted 2014-11-26; First posted 2014-12-03 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hypophosphatasia (HPP)
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

SUMMARY:
In this prospective, observational, long term registry patients of all ages with a diagnosis of hypophosphatasia (HPP) are followed at participating sites in multiple countries.

DETAILED DESCRIPTION:
The HPP Registry is an observational, prospective, long-term registry designed to collect data on HPP epidemiology, disease history, clinical course, symptoms and burden of disease from patients of all ages who have a diagnosis of HPP.

Evaluation of safety and effectiveness data in patients with HPP who have/are receiving treatment with Asfotase alfa

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, of any age, with a confirmed diagnosis of HPP.
* Participant must have documented alkaline phosphatase (ALP) activity below the lower limit of normal for age and sex, or a documented ALPL gene mutation.
* Participant or legal representative is able to read and/or understand the informed consent and study questionnaires in the local language.
* Signed informed consent and medical records release by the patient or legal representative. Patient or patient's parent/legal representative must be willing and able to give written informed consent, and the patient must be willing to give written informed assent, if appropriate and required by local regulations.

Exclusion Criteria:

* Currently participating in an Alexion-sponsored clinical trial. Enrollment in the Registry will not exclude a patient from enrolling in a future clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hypophosphatasia (HPP)
Sampling Method: Probability Sample
Enrollment: 1571 (Estimated)
Dates: Start 2015-01-20 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Natural History Information | 1 Year
  To collect information on the natural history of HPP from patients of all ages, including pediatric patients and adults with HPP, regardless of age at onset.
Burden of Disease/Patient-reported Outcomes | 1 year
  Age-appropriate PRO data will be collected using instruments to asses below: Pain, Motor Capacity, Functional Status/Disability, including Activities of Daily Living (ADL), Quality of Life (QoL)
Characterize the epidemiology of the HPP population. | 1 year
  To characterize the epidemiology of the HPP population. Inclusion of all classifications of HPP is planned: pediatric-onset (perinatal-, infantile-, and juvenile-onset), adult-onset, benign perinatal, and odontohypophosphatasia.
Long-Term Safety and Effectiveness of Asfotase Alfa | 1 year
  To collect and evaluate long-term safety and effectiveness data in HPP patients who have/are receiving treatment with asfotase alfa.

CONTACTS AND LOCATIONS:
Locations (64):
- United States (19):
  - Research Site, Centennial, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Tampa, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, Mineola, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Madison, Wisconsin
- Australia (4):
  - Research Site, Clayton, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Herston
  - Research Site, South Brisbane
- Research Site, Linz, Austria
- Canada (4):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Oakville, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- France (7):
  - Research Site, Toulouse, Haute Garonne
  - Research Site, Lille, Nord
  - Research Site, Paris, Paris
  - Research Site, Poitiers, Vienne
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Le Kremlin-Bicêtre, Île-de-France Region
- Germany (10):
  - Research Site, Bad Reichenhall, Bavaria
  - Research Site, Würzburg, Bavaria
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Dresden, Saxony
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Giessen
  - Research Site, Homburg
  - Research Site, Mainz
- Italy (5):
  - Research Site, Milan, Milano
  - Research Site, Florence
  - Research Site, Pisa
  - Research Site, Rome
  - Research Site, San Giovanni Rotondo
- Poland (2):
  - Research Site, Lodz
  - Research Site, Warsaw
- Research Site, Riyadh, Saudi Arabia
- Research Site, Madrid, Spain
- United Kingdom (10):
  - Research Site, Bristol, Avon
  - Research Site, London, Greater London
  - Research Site, Leicester, Leicestershire
  - Research Site, Stanmore, Middlesex
  - Research Site, Oxford, Oxfordshire
  - Research Site, Sheffield, South Yorkshire
  - Research Site, Dundee, Tayside Region
  - Research Site, Newcastle upon Tyne, Tyne & Wear
  - Research Site, Birmingham, West Midlands
  - Research Site, Belfast

REFERENCES:
- [Background] Dahir KM, Seefried L, Kishnani PS, Petryk A, Hogler W, Linglart A, Martos-Moreno GA, Ozono K, Fang S, Rockman-Greenberg C. Clinical profiles of treated and untreated adults with hypophosphatasia in the Global HPP Registry. Orphanet J Rare Dis. 2022 Jul 19;17(1):277. doi: 10.1186/s13023-022-02393-8. PMID 35854311
- [Background] Dahir KM, Kishnani PS, Martos-Moreno GA, Linglart A, Petryk A, Rockman-Greenberg C, Martel SE, Ozono K, Hogler W, Seefried L. Impact of muscular symptoms and/or pain on disease characteristics, disability, and quality of life in adult patients with hypophosphatasia: A cross-sectional analysis from the Global HPP Registry. Front Endocrinol (Lausanne). 2023 Mar 27;14:1138599. doi: 10.3389/fendo.2023.1138599. eCollection 2023. PMID 37051203
- [Background] Hogler W, Linglart A, Petryk A, Kishnani PS, Seefried L, Fang S, Rockman-Greenberg C, Ozono K, Dahir K, Martos-Moreno GA. Growth and disease burden in children with hypophosphatasia. Endocr Connect. 2023 Apr 25;12(5):e220240. doi: 10.1530/EC-22-0240. Print 2023 May 1. PMID 36917043
- [Background] Hogler W, Langman C, Gomes da Silva H, Fang S, Linglart A, Ozono K, Petryk A, Rockman-Greenberg C, Seefried L, Kishnani PS. Diagnostic delay is common among patients with hypophosphatasia: initial findings from a longitudinal, prospective, global registry. BMC Musculoskelet Disord. 2019 Feb 14;20(1):80. doi: 10.1186/s12891-019-2420-8. PMID 30764793
- [Background] Kishnani PS, Martos-Moreno GA, Linglart A, Petryk A, Messali A, Fang S, Rockman-Greenberg C, Ozono K, Hogler W, Seefried L, Dahir KM. Effectiveness of asfotase alfa for treatment of adults with hypophosphatasia: results from a global registry. Orphanet J Rare Dis. 2024 Mar 8;19(1):109. doi: 10.1186/s13023-024-03048-6. PMID 38459585
- [Background] Martos-Moreno GA, Rockman-Greenberg C, Ozono K, Petryk A, Kishnani PS, Dahir KM, Seefried L, Fang S, Hogler W, Linglart A. Clinical Profiles of Children with Hypophosphatasia prior to Treatment with Enzyme Replacement Therapy: An Observational Analysis from the Global HPP Registry. Horm Res Paediatr. 2024;97(3):233-242. doi: 10.1159/000531865. Epub 2023 Jul 13. PMID 37442110
- [Background] Seefried L, Dahir K, Petryk A, Hogler W, Linglart A, Martos-Moreno GA, Ozono K, Fang S, Rockman-Greenberg C, Kishnani PS. Burden of Illness in Adults With Hypophosphatasia: Data From the Global Hypophosphatasia Patient Registry. J Bone Miner Res. 2020 Nov;35(11):2171-2178. doi: 10.1002/jbmr.4130. Epub 2020 Aug 10. PMID 32654183
- [Background] Kishnani PS, Seefried L, Dahir KM, Martos-Moreno GA, Linglart A, Petryk A, Mowrey WR, Fang S, Ozono K, Hogler W, Rockman-Greenberg C. New insights into the landscape of ALPL gene variants in patients with hypophosphatasia from the Global HPP Registry. Am J Med Genet A. 2024 Nov;194(11):e63781. doi: 10.1002/ajmg.a.63781. Epub 2024 Jun 17. PMID 38884565
- [Background] Kishnani PS, Seefried L, Dahir KM, Martos-Moreno GA, Hogler W, Greenberg CR, Fang S, Petryk A, Mowrey WR, Linglart A, Ozono K. Disease burden by ALPL variant number in patients with non-life-threatening hypophosphatasia in the Global HPP Registry. J Med Genet. 2025 Mar 20;62(4):249-257. doi: 10.1136/jmg-2024-110383. PMID 39965917
- [Background] Tornero C, Martos-Moreno GA, Guanabens N, Florez H, Ribera A, Aguado P. Clinical characterization and impact of hypophosphatasia in Spain: An observational analysis of the Spanish cohort included in the Global HPP Registry. Med Clin (Barc). 2025 Nov;165(5):107120. doi: 10.1016/j.medcli.2025.107120. Epub 2025 Jul 25. English, Spanish. PMID 40714462
- [Background] Kishnani PS, Seefried L, Ozono K, Martos-Moreno GA, Rockman-Greenberg C, Fowler D, Burke LK, Mowrey WR, Rush ET, Ebeling PR, Hogler W, Linglart A, Fang S, Petryk A, Dahir KM. The Global Hypophosphatasia Registry: lessons learned from a decade of real-world data. Orphanet J Rare Dis. 2025 Nov 24;20(1):626. doi: 10.1186/s13023-025-04129-w. PMID 41286962